CLINICAL TRIAL: NCT06106711
Title: The Impact of Adverse Events, Produced by Antibodies Conjugates, on Quality of Life in Patients With Metastatic Breast Cancer: Multicentric, Observational Study (EVA).
Acronym: EVA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-22
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study stems from the need to detect adverse events arising after the administration of Antibody-Drug Conjugates (ADCs) used in the treatment of metastatic breast cancer in a real life context and to correlate the same with the quality of life reported by patients.

DETAILED DESCRIPTION:
The study stems from the need to detect adverse events arising after the administration of ADCs used in the treatment of metastatic breast cancer in a real life context and to correlate the same with the quality of life reported by patients.Through the findings of toxicities related to the ADCs, it will be possible to highlight which are the issues that most affect patients undergoing these cancer treatments. The analysis of the data collected will also make it possible to highlight any toxicities not yet considered or/and of new onset. In addition useful elements may emerge from responses to the quality of life questionnaire, to cope with the difficulties expressed by patients regarding daily life activities, social relations, work and family. Such contributions will be fundamental to the construction of integrated care pathways, the aim of which is to involve a specialized nurse as part of a multidisciplinary team.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Age ≥ 18 years;
* Signature of consent to participate in the study and to the processing of personal data (Privacy);
* Diagnosis of stage IV breast cancer;
* Systemic treatment with T-DM1, T-DXD or SG as monotherapy;
* Absence of cognitive decline, expressed by a score greater than or equal to 4 on the Six Item Screener questionnaire;
* Good understanding of the Italian language;
* Willingness and ability to adhere to scheduled visits, treatment plan, laboratory tests and study procedures.

Exclusion Criteria:

* All patients who do not meet the above criteria will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 92 patients diagnosed with stage IV breast cancer treated at the Department of Medical Oncology and Cancer Prevention, IRCCS National Cancer Institute of Aviano and at the other involved clinical centers considered eligible for the study will be enrolled, after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) arising during treatment and degree of toxicity | up to 1 year
  Frequency adverse events (AEs) arising during treatment with TDM-1, T-DXd and SG
Adverse events (AEs) arising during treatment and degree of toxicity | up to 1 year
  description of degree of toxicity of AEs classified using the international classification system CTCAE (version 5.0)
Quality of life of patients during treatment | up to 1 year
  To assess the quality of life of patients treated with TDM-1, T-DXd, and SG through the administration of the EORTC QLQ-C30 questionnaire. Results will be reported as median and quartiles

SECONDARY OUTCOMES:
Dose-reduction | up to 1 year
  to identify the percentage of patients who require a reduction in dosage due to suboptimal treatment tolerance
Treatment discontinuation | up to 1 year
  Identify the percentage of patients who discontinues cancer therapy due to suboptimal treatment tolerance
AEs - level of distress | up to 1 year
  difference in distress levels measured with Distress thermometer between patients with different AEs secondary to cancer treatments
To describe the actions taken to manage treatment-related AEs | up to 1 year
  Description of the actions taken to manage treatment-related AEs
Analyze the level of concordance between the AEs detected by health care personnel and the patient's subjective assessment | up to 1 year
  Concordance between the AEs detected by health care personnel and the patient's subjective assessment
Sources of distress | up to 1 year
  Frequency for answers to Distress thermometer problem list

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Mazzega Fabbro, MSc, Principal Investigator — Centro di Riferimento Oncologico (CRO), IRCCS
Locations (3):
- Italy (3):
  - Centro di Riferimento Oncologico (CRO), Aviano, Pordenone
  - Fondazione IRCCS Istituto Nazionale dei tumori, Milan
  - Istituto Nazionale Tumori IRCCS G. Pascale, Napoli